CLINICAL TRIAL: NCT01312090
Title: Chronic Intermittent Cold Exposure on Weight Loss
Acronym: CICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Sanna Kaye, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PS09RUSRAS; T1070RUSRA (Other: Helsinki University Central Hospital registry)
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: Weight loss; brown adipose tissue; white adipose tissue; muscle, metabolism; cold exposure
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Counseling; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional weight loss treatment group (Active Comparator): Eating and physical activity counseling and behavioral therapy for weight loss.
  Interventions: Behavioral: counseling and behavioral therapy for weight loss
- Cryo group (Experimental): Eating and physical activity counseling and behavioral therapy for weight loss will be provided to all subjects.
  The subjects in the cryo group will be given whole-body cryotherapy 1-3 times a week for the 4-month-treatment period
  Interventions: Biological: Whole body cryotherapy

INTERVENTIONS:
Biological: Whole body cryotherapy — Cryotherapy: The whole-cody cryotherapy device (Univers Cryo-Combi;Oy MJG Univers Ab, Helsinki, Finland) consists of 3 chambers set at different temperatures. The first 2 chambers are meant for precooling (-30°Cand-60°C), and the patient remains in these for a very short time. The third chamber temperature reaches -110°C, and the patient remains inside for 3-4 minutes wearing a bathing suit or trunks, acral parts covered.
  Arms: Cryo group
Behavioral: counseling and behavioral therapy for weight loss — Weight loss intervention with Very Low Calory Diet (VLCD, 500-1000 kcal / d + dietary supplements) and group and individual treatment (eating, physical activity counseling and behavioural therapy).
  Arms: Conventional weight loss treatment group

SUMMARY:
1. To test whether chronic intermittent cold exposure is more effective in programmed body weight loss when compared to conventional programmed weight loss.
2. To measure the metabolic responses (e.g. in the white and brown adipose tissue, muscle and circulating markers) of treatment with chronic intermittent cold exposure and conventional treatment
3. To measure tissue specific changes of weight loss and the treatment with chronic intermittent cold exposure in glucose uptake rate in adipose organ (white and brown adipose tissue), liver, myocardium, skeletal muscle and brain
4. To measure tissue specific biochemical indicators before and after treatment with chronic intermittent cold exposure from white adipose tissue and skeletal muscle.
5. To compare changes in body composition and fat distribution after weight loss using chronic cold exposure or using conventional method

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 (inclusive)
* Body weight less than 120 kg
* Weight stability for 3 months
* Plasma triglyceride concentration less than 3.0 mmol/l
* Plasma HDL-cholesterol more than 0.9 mmol/l in males and more than 1.0 mmol/l in females
* Blood pressure less than 140/90 mmHg (inclusive)
* Normal glucose tolerance or impaired glucose tolerance but not diabetes (fasting glucose < 7.0 mmol/l or 2 h glucose in the oral glucose tolerance test < 11.1 mmol/l)

Exclusion Criteria:

* Smoking
* Frequent weight loss attempts
* Pregnancy or lactation
* Diabetes mellitus
* Hypo/hyperthyreosis
* Cardiovascular disease, stroke or neurological disorder
* Medication (antihypertensive and antidiabetic drugs, lipid lowering drugs, antidepressants, corticosteroids)
* Claustrophobia
* Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results.
* Presence of any ferromagnetic objects that would make MRI imaging contraindicated

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
weight loss | looking forward using periodic observations collected predominantly during 12 months following subject enrollment
  Effect of chronic intermittent cold exposure and conventional treatment on weight loss

SECONDARY OUTCOMES:
Glucose uptake | 4 months from admission
  Effect of chronic intermittent cold exposure and conventional treatment on glucose uptake of brown and white adipose tissue, liver, myocardium, skeletal muscle and brain (PET-scan).
energy metabolism | 12 months from admission
  Effect of chronic intermittent cold exposure and conventional treatment on energy metabolism
behavioural patterns | 12 months from admission
  Effect of chronic intermittent cold exposure and conventional treatment on behavioural patterns
muscle metabolism | 12 months from admission
  Effect of chronic intermittent cold exposure and conventional treatment on muscle metabolism
white adipose tissue metabolism | 12 months from admission
  Effect of chronic intermittent cold exposure and conventional treatment on white adipose tissue metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi H Pietilainen, MD, PhD, Principal Investigator — Obesity research Unit, Department of Medicine, Helsinki University Central Hospital

REFERENCES:
- [Derived] van der Kolk BW, Heinonen S, White JW, Wagner A, Karppinen JE, Saari S, Muniandy M, Metsikko S, Dillon ET, Groop PH, Saarinen T, Le Roux CW, Virtanen KA, Docherty NG, Pirinen E, Juuti A, Pietilainen KH. Human Skeletal Muscle Mitochondria Responses to Weight Loss Induced by Bariatric Surgery or Lifestyle Intervention. Acta Physiol (Oxf). 2026 Feb;242(2):e70150. doi: 10.1111/apha.70150. PMID 41507695
- [Derived] Karppinen JE, Suojanen L, Heinonen S, Kaye S, van der Kolk BW, White JW, Orava J, Lee SHT, Dillon E, Muniandy M, Rissanen A, le Roux CW, Docherty N, Pajukanta P, Virtanen KA, Pietilainen KH. Effects of Whole-Body Cryotherapy Combined With Conventional Obesity Management Versus Obesity Management Alone: A Clinical Trial. Obesity (Silver Spring). 2025 Nov;33(11):2112-2127. doi: 10.1002/oby.70019. Epub 2025 Sep 3. PMID 40903800
- [Derived] van der Kolk BW, Muniandy M, Kaminska D, Alvarez M, Ko A, Miao Z, Valsesia A, Langin D, Vaittinen M, Paakkonen M, Jokinen R, Kaye S, Heinonen S, Virtanen KA, Andersson DP, Mannisto V, Saris WH, Astrup A, Ryden M, Blaak EE, Pajukanta P, Pihlajamaki J, Pietilainen KH. Differential Mitochondrial Gene Expression in Adipose Tissue Following Weight Loss Induced by Diet or Bariatric Surgery. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1312-1324. doi: 10.1210/clinem/dgab072. PMID 33560372